CLINICAL TRIAL: NCT00003243
Title: A Phase I Trial of Combined Chemotherapy and Donor Lymphocyte Infusion for Aggressive Hematologic Malignancies in Relapse After Allogeneic Bone Marrow Transplantation
Brief Title: Combination Chemotherapy Plus Infusion of White Blood Cells in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066119, J9743; P30CA006973 (NIH); JHOC-97112101; NCI-V98-1387
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; acute undifferentiated leukemia; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; secondary acute myeloid leukemia; previously treated myelodysplastic syndromes; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Biphenotypic, Acute; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — aldesleukin; Filgrastim; Cyclophosphamide; Etoposide

INTERVENTIONS:
Biological: aldesleukin
Biological: filgrastim
Biological: therapeutic allogeneic lymphocytes
Drug: cyclophosphamide
Drug: etoposide
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. White blood cells from donors may be able to kill cancer cells in patients who have hematologic cancer that has recurred following bone marrow transplantation.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy plus infusion of donated white blood cells in treating patients who have hematologic cancer that has recurred after bone marrow transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of doxorubicin HCl liposome when combined with etoposide, cyclophosphamide, and allogeneic donor lymphocyte infusion with or without interleukin-2 after allogeneic bone marrow transplantation in patients with relapsed or persistent aggressive hematologic malignancies.

OUTLINE: This is a partially randomized, dose-escalation study of doxorubicin HCl liposome (LipoDox).

Patients enter 1 of 4 cohorts.

* Cohort 1: Three to six patients receive induction comprising etoposide IV over 1 hour on days 1-3, cyclophosphamide IV over 1-2 hours on day 8, and allogeneic donor lymphocyte infusion on day 10. Filgrastim (G-CSF) is administered subcutaneously (SC) or IV daily beginning on day 10 and continuing until blood counts recover.
* Cohort 2: In the absence of dose-limiting toxicity (DLT) on cohort 1, 3-6 patients receive treatment as in cohort 1 and LipoDox IV over 2 hours on day 1.
* Cohort 3: In the absence of DLT on cohort 2, 3-6 patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive treatment as in cohort 1 plus a higher dose of LipoDox IV over 2 hours on day 1.
  * Arm II: Patients receive treatment as in cohort 1 and interleukin-2 (IL-2) SC on days 10-12.

If DLT is reached on cohort 2, 3-6 patients receive treatment as in arm II.

* Cohort 4: In the absence of DLT on arms I and II, patients receive treatment as in cohort 1, LipoDox as in arm I, and IL-2 as in arm II.

Cohorts of 3-6 patients receive escalating doses of LipoDox until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience DLT.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 12-15 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of relapsed or persistent acute leukemia, myelodysplasia, aggressive non-Hodgkin's lymphoma (NHL), or chronic myeloid leukemia in transformed phase (accelerated phase or blast crisis) after allogeneic bone marrow transplantation (BMT)
* Aggressive NHL defined as diffuse mixed, diffuse large cell, diffuse small noncleaved cell, and lymphoblastic histologies
* No active acute graft versus host disease (GVHD) or extensive chronic GVHD

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* More than 4 weeks

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No severe psychiatric illness or mental deficiencies

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 6 months since prior allogeneic BMT
* No other concurrent interleukin-2
* No other concurrent immunomodulatory medication (e.g., interferon)

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent steroids

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent immunosuppressive medication (e.g., cyclosporine) for GVHD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-01

CONTACTS AND LOCATIONS:
Overall Officials: Ephraim J. Fuchs, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States